CLINICAL TRIAL: NCT05843448
Title: Pilot Study of an IDO and PD-L1 Peptide Based Immune-Modulatory Therapeutic (IO102-IO103) in Combination With Pembrolizumab for BCG-Unresponsive or Intolerant, Non-Muscle Invasive Bladder Cancer
Brief Title: IDO and PD-L1 Peptide Based Immune-Modulatory Therapeutic (IO102-IO103) in Combination With Pembrolizumab for BCG-Unresponsive or Intolerant, Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: IO Biotech (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mamta Parikh, Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#290; NCI-2023-02851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#290 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: High Risk Non-Muscle Invasive Bladder Urothelial Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (IO102-IO103, pembrolizumab) (Experimental): Patients receive PD-L1/IDO peptide vaccine SC and pembrolizumab IV on study. Patients also undergo CT and/or CT/PET and collection of blood samples throughout the trial.
  Interventions: Biological: PD-L1/IDO Peptide Vaccine; Biological: Pembrolizumab

INTERVENTIONS:
Biological: PD-L1/IDO Peptide Vaccine — Given SC
  Other Names: IO102-IO103 Peptide Vaccine; IO103/IO102 Peptide Vaccine; PD-L1/IDO Peptide
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial tests the safety and side effects of a PD-L1/IDO peptide vaccine (IO102-IO103) in combination with pembrolizumab in treating patients with non-muscle invasive bladder cancer. IO102-IO103 is a novel IDO and PD-L1 peptide based immune-modulatory therapeutic. It is designed to activate the patient's own immune cells (called T-cells) to fight the tumor and stop the tumor cells escaping from the body's immune system. IO102-IO103 works to directly kill tumor cells and remove the body's immune suppressive cells, which are cells that prevent the immune system from fighting the tumor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving IO102-IO103 in combination with pembrolizumab may make tumor cells more visible/recognizable to the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: I. Evaluate the feasibility, safety and toxicity of the PD-L1/IDO peptide vaccine (IO102-IO103) in combination with pembrolizumab in patients with Bacillus Calmette-Guerin (BCG)-unresponsive or intolerant, non-muscle invasive bladder cancer (NMIBC).

SECONDARY OBJECTIVES: I. To assess preliminary efficacy of IO102-IO103 in combination with pembrolizumab. II. To obtain preliminary efficacy of IO102-IO103 in combination with pembrolizumab.

OUTLINE: Patients receive PD-L1/IDO peptide vaccine subcutaneously (SC) and pembrolizumab intravenously (IV) on study. Patients also undergo computed tomography (CT) and/or CT/positron emission tomography (PET) and collection of blood samples throughout the trial.After completion of study treatment, patients are followed up for 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years of age
* Histologically confirmed high-risk NMIBC (T1, high-grade Ta, or carcinoma in situ [CIS]/Tis). Mixed histologies are allowed if predominantly transitional cell histology. Archival tissue or planned cystoscopy within 28 day of planned initiation of treatment
* Maximally resected tumor on study entry
* Cystectomy ineligible or declined
* Two induction courses of BCG attempted, regardless of exact doses received
* ECOG (Eastern Cooperative Oncology Group) performance status score of 0 - 2
* Life expectancy >= 6 months
* Absolute neutrophil count (ANC) > 1000 cells/uL (=< 14 days of the first study treatment)
* Platelet count > 50,000/uL (=< 14 days of the first study treatment)
* Hemoglobin > 8 g/dL (=< 14 days of the first study treatment)
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 5 x upper limit of normal (ULN) (=< 14 days of the first study treatment)
* Alkaline phosphatase =< 5 x upper limit of normal (ULN) (=< 14 days of the first study treatment)
* Total bilirubin =< 2 x ULN (=< 14 days of the first study treatment)
* Creatinine clearance > 30 mL/min as measured using Cockcroft-Gault equation or the estimated glomerular filtration rate from the Modification of Diet in Renal Disease Study (=< 14 days of the first study treatment)
* International normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless the subject is receiving anticoagulant therapy. Individuals on anticoagulant therapy should have a prothrombin time (PT) or partial thromboplastin time (PTT) within therapeutic range of intended use and no history of severe hemorrhage
* Ability to understand and willingness to sign an informed consent document
* Ability to adhere to the study visit schedule and other protocol requirements
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use methods of contraception

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment may, in the opinion of the investigator, have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the patient's safety or compliance on trial
* Known history of positive test for human immunodeficiency virus (HIV) with CD4 < 200 or acquired immunodeficiency syndrome (AIDS)-defining condition
* Known active tuberculosis
* Active infection requiring systemic therapy, including active or intractable urinary tract infection (UTI)
* Previous treatment with checkpoint inhibitors targeting either PD-(L)1 or CTLA-4
* Prior exposure to IO102 or IO103
* Received systemic chemotherapy, targeted small molecule therapy, or radiotherapy =< 2 weeks before study treatment initiation
* Any adverse events from prior cancer therapy have resolved to grade =< 1 according to Common Terminology Criteria for Adverse Events (CTCAE) version 5
* Congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis
* Any medical condition requiring systemic steroid equivalent to prednisone > 10 mg daily or immunosuppressive therapy within 14 days or 5 half-lives prior to first dose of trial therapy. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible. Patients who have adrenal insufficiency and hypophysitis from prior immunotherapy if they are on stable medical replacement doses are eligible
* Received a live or live-attenuated vaccine =< 30 days before the first dose of study treatment. Administration of killed vaccines, messenger ribonucleic acid (mRNA) based vaccines (e.g., COVID-19), and vector based vaccines are allowed
* Pregnant and/or breast feeding women. If a urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required =< 24 hours prior to planned treatment initiation
* Evidence of active interstitial lung disease or history of non-infectious pneumonitis requiring systemic steroids
* Known allergy or reaction to any component of either study drug formulation
* Any condition that would prohibit the understanding or rendering of informed consent
* Any condition that in the opinion of the investigator would interfere with the patient's safety or compliance while on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose
  Safety and toxicity will be evaluated according to Common Terminology Criteria for Adverse Events version 5.0 and pre-defined treatment-limiting toxicities.

SECONDARY OUTCOMES:
Complete response (CR) | At 3 months
  The CR rate will be estimated as the proportion of participants who experience an objective response, along with its exact 95% confidence interval. The CR rate at 3 months will be used to determine whether the trial will be expanded based on Simon's two-stage design.
Event-free survival | At 18 months
  Kaplan-Meier methods will be used to estimate event-free (including recurrence on biopsy, development of muscle-invasive urothelial carcinoma, progression requiring radical cystectomy, or development of metastatic disease) survival at 18 months, along with 95% confidence intervals.
Cystectomy-free survival | At 18 months
  Kaplan-Meier methods will also be used to estimate cystectomy-free survival at 18 months, along with 95% confidence intervals.
Duration of response (DOR) | Up to 3 years
  DOR will be analyzed using Kaplan-Meier methods; medians and 95% confidence intervals will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States